CLINICAL TRIAL: NCT00990990
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled Study To Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of PNU-100480 (PF-02341272) After Administration Of Multiple Escalating Oral Doses To Healthy Adult Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics And Measurement Of Whole Blood Activity (WBA) Of PNU-100480 After Multiple Oral Doses In Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sequella, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: B1171002
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Tuberculosis
Keywords: Safety tolerability pharmacokinetics (PK) pharmacodynamics whole blood activity (WBA) PNU-100480 linezolid pyrazinamide multiple dose
MeSH Terms: conditions — Tuberculosis | interventions — PNU-100480; Linezolid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Cohort 1 (Experimental)
  Interventions: Drug: PNU-100480; Drug: Placebo
- Cohort 2 (Experimental)
  Interventions: Drug: PNU-100480; Drug: Placebo
- Cohort 3 (Experimental)
  Interventions: Drug: PNU-100480; Drug: Placebo
- Cohort 4 (Experimental)
  Interventions: Drug: PNU-100480; Drug: Placebo
- Cohort 5 (Experimental)
  Interventions: Drug: PNU-100480; Drug: Placebo
- Cohort 6 (optional) (Experimental)
  Interventions: Drug: PNU-100480; Drug: Placebo
- Linezolid Cohort (Experimental)
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: PNU-100480 — 100 mg BID for 14 days
  Arms: Cohort 1
Drug: Placebo — to match 100 mg BID for 14 days
  Arms: Cohort 1
Drug: PNU-100480 — 300 mg BID for 14 days
  Arms: Cohort 2
Drug: Placebo — to match 300 mg BID for 14 days
  Arms: Cohort 2
Drug: PNU-100480 — 600 mg BID for 14 days
  Arms: Cohort 3
Drug: Placebo — to match 600 mg BID for 14 days
  Arms: Cohort 3
Drug: PNU-100480 — 1200 mg QD for 14 days
  Arms: Cohort 4
Drug: Placebo — to match 1200 mg QD for 14 days
  Arms: Cohort 4
Drug: PNU-100480 — 600 mg BID for 28 days with pyrazinamide (25 mg/kg up to 2 g) QD on Days 27-28
  Arms: Cohort 5
Drug: Placebo — placebo to match 600 mg BID for 28 days with pyrazinamide (25 mg/kg up to 2 g) QD on Days 27-28
  Arms: Cohort 5
Drug: PNU-100480 — PNU-100480 dose up to total of 1200 mg daily for 28 days with pyrazinamide (25 mg/kg up to 2 g) QD on Days 27-28
  Arms: Cohort 6 (optional)
Drug: Placebo — placebo to match dose up to total of 1200 mg daily for 28 days with pyrazinamide (25 mg/kg up to 2 g) QD on Days 27-28
  Arms: Cohort 6 (optional)
Drug: Linezolid — 300 mg QD for 4 days (open label)
  Arms: Linezolid Cohort

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics of multiple doses of PNU-100480 given for 14 or 28 days. Killing activity against the bacterium that causes tuberculosis (TB) will also be measured. The effect of adding an additional tuberculosis (TB) agent (given for 2 days) in addition to PNU-100480 will be evaluated. Linezolid open label to determine activity in whole blood assay (WBA).

DETAILED DESCRIPTION:
Evaluate safety, tolerability, pharmacokinetics and whole blood activity (WBA) of PNU-100480 given for 14 or 28 days; evaluate WBA of PNU with pyrazinamide; evaluate WBA of linezolid

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers willing and able to be confined to the Clinical Research Unit and comply with study schedule.
* Women of non-childbearing potential only.

Exclusion Criteria:

* History of hypersensitivity to, or intolerance of, linezolid.
* Antibiotic treatment within 14 days prior to dosing, or any previous antibiotic use at the discretion of the investigator.
* Previous history of irritable bowel syndrome (IBS) or inflammatory bowel disease (IBD).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of ascending oral doses of PNU-100480 administered as extemporaneously prepared suspension (EPS) over 14 and 28 days in healthy adult volunteers. | Monitor adverse events daily; safety eval pre-dose, specified times , discharge, follow-up/as needed

SECONDARY OUTCOMES:
To characterize the single dose and steady state pharmacokinetics of ascending oral doses of PNU-100480 administered over 14 and 28 days in healthy adult volunteers with regard to the parent drug and its metabolites. | Full and sparse PK sampling from Day 1 through final day of dosing
To characterize the bactericidal activity in blood of orally administered PNU-100480 against intracellular M. tuberculosis in relation to blood concentrations ofPNU-100480 and its metabolites. | Full and sparse sampling from Day 1 through final day of dosing
To characterize the effect of once a day administration of pyrazinamide for 2 days on the pharmacokinetics and bactericidal activity in blood of orally administered PNU-100480 against intracellular M. tuberculosis (Cohorts 5 and 6, Days 27-28 only). | Days 27-28 as applicable
To characterize pharmacokinetics and bactericidal activity in blood of orally administered linezolid against intracellular M. tuberculosis following 4 days of QD dosing. | As applicable up to Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Beth Ferstenberg, M.D., Study Director — Sequella, Inc.
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Wallis RS, Jakubiec WM, Kumar V, Silvia AM, Paige D, Dimitrova D, Li X, Ladutko L, Campbell S, Friedland G, Mitton-Fry M, Miller PF. Pharmacokinetics and whole-blood bactericidal activity against Mycobacterium tuberculosis of single doses of PNU-100480 in healthy volunteers. J Infect Dis. 2010 Sep 1;202(5):745-51. doi: 10.1086/655471. PMID 20629533
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1171002&StudyName=Safety%2C%20Tolerability%2C%20Pharmacokinetics%20And%20Measurement%20Of%20Whole%20Blood%20Activity%20%28WBA%29%20Of%20PNU-100480%20After%20Multiple%20Oral%20Doses%20In%20Heal